CLINICAL TRIAL: NCT00420199
Title: A Phase IIIB Multicenter, Randomized, Double-Blind, Placebo-controlled Study to Assess Short-term Changes in Synovitis and Structural Damage Outcomes in Subjects With Active Rheumatoid Arthritis and Inadequate Response to Methotrexate, Treated With Abatacept Versus Placebo on a Background Therapy With Methotrexate
Brief Title: A Phase IIIb Study of BMS-188667 in Subjects With Active Rheumatoid Arthritis and Inadequate Response to Methotrexate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM101-119; Eudract: 2006-003768-67
Record Dates: First submitted 2007-01-08; First posted 2007-01-09 (Estimated); Results first posted 2011-05-17 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Active Rheumatoid Arthritis
MeSH Terms: interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Abatacept + Methotrexate (Double-blind period) (Active Comparator)
  Interventions: Drug: Abatacept
- Placebo + Methotrexate (Double-blind period) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Abatacept — Vials (250 mg/vial), intravenous (IV), 10 mg/kg, monthly infusion , 12 months of treatment
  Other Names: (BMS-188667); Orencia
  Arms: Abatacept + Methotrexate (Double-blind period)
Drug: Placebo — Intravenous (IV) bags, IV, 0 mg, monthly infusion, 12 months of treatment
  Arms: Placebo + Methotrexate (Double-blind period)

SUMMARY:
The only trial in participants who are methotrexate-inadequate responders and have active Rheumatoid Arthritis, in which gadolinium-enhanced Magnetic Resonance Imaging; Bone Mineral Density; and biochemical markers of bone, cartilage, and synovial tissue metabolism are used to evaluate early effects (4 months) of Abatacept on inflammation/structural damage. Study will provide valuable mechanism-of-action information on how Abatacept exerts its effects (including on bone) through new techniques.

ELIGIBILITY:
Inclusion Criteria:

* Disease activity as defined by a Disease Activity Score 28-C-Reactive Protein (CRP) >3.2 or >6 swollen and ≥6 tender joints and CRP greater than the upper limit of normal
* At least 1 erosion in hands/wrists or positive anticyclic citrullinated peptides or rheumatoid factor
* Clinically detectable synovitis of at least 1 wrist/ankle at screening and baseline
* Participants must have been treated with methotrexate, on a weekly dose of at least 15 mg or a maximum tolerated dose (such as, 10 mg weekly) for at least 3 months before screening. Dose of methotrexate must be stable for at least 28 days prior to the first study dose (Day 1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-05; Primary Completion 2009-08 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (8):
- Belgium (2):
  - Local Institution, Brussels
  - Local Institution, Yvoir
- Local Institution, Berlin, Germany
- Local Institution, Amsterdam, Netherlands
- Local Institution, Barcelona, Spain
- Local Institution, Stockholm, Sweden
- United Kingdom (2):
  - Local Institution, London, Greater London
  - Local Institution, Leeds, North Yorkshire

REFERENCES:
- [Derived] Conaghan PG, Durez P, Alten RE, Burmester GR, Tak PP, Klareskog L, Catrina AI, DiCarlo J, Gaillez C, Le Bars M, Zhou X, Peterfy C. Impact of intravenous abatacept on synovitis, osteitis and structural damage in patients with rheumatoid arthritis and an inadequate response to methotrexate: the ASSET randomised controlled trial. Ann Rheum Dis. 2013 Aug;72(8):1287-94. doi: 10.1136/annrheumdis-2012-201611. Epub 2012 Aug 21. PMID 22915624
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Groups:
- Abatacept (ABA) + Methotrexate (MTX): Abatacept was administered intravenously (IV) on Day 1, 15, 29 and every 28 days up to and including Day 113.Abatacept was given as a dose based on body weight: 500 mg for participants weighing < 60 kg, 750 mg for participants weighing 60 to 100 kg and 1 gram for participants weighing > 100 kg.
- Placebo (PLA) + MTX: PLA was administered IV on Day 1, 15, 29 and every 28 days up to and including Day 113. In addition, participants received a weekly dose of MTX of at least 15 mg or a maximum tolerated dose (ie, 10 mg weekly)
Period: Overall Study
Arm/Group | Abatacept (ABA) + Methotrexate (MTX) | Placebo (PLA) + MTX
Started | 27 | 23
Completed | 26 | 23
Not Completed | 1 | 0
Not completed — Participant no longer met study criteria | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Abatacept (ABA) + Methotrexate (MTX): Abatacept was administered IV on Day 1, 15, 29 and every 28 days up to and including Day 113.Abatacept was given as a dose based on body weight: 500 mg for participants weighing < 60 kg, 750 mg for participants weighing 60 to 100 kg and 1 gram for participants weighing > 100 kg.
- Total: Total of all reporting groups
Arm/Group | Abatacept (ABA) + Methotrexate (MTX) | Placebo (PLA) + MTX | Total
Number analyzed (Participants) | 27 | 23 | 50
Age Continuous [Mean (Standard Deviation); unit: years] | 51.7 (11.2) | 52.5 (11.5) | 52.1 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 11 | 7 | 18
Region of Enrollment [Number; unit: participants]
  Belgium | 9 | 7 | 16
  Germany | 10 | 6 | 16
  Netherlands | 3 | 4 | 7
  Spain | 2 | 2 | 4
  Sweden | 2 | 3 | 5
  United Kingdom | 1 | 1 | 2
Rheumatoid Factor (RF) Status [Number; unit: participants] — Rheumatoid factor (RF or RhF) is an autoantibody (antibody directed against an organism's own tissues) most relevant in rheumatoid arthritis. It is an antibody against the Fc portion of Immunoglobulin (Ig)G, which is itself an antibody. RF and IgG join to form immune complexes which contribute to the disease process.
  participants
    Negative | 12 | 4 | 16
    Positive | 15 | 19 | 34
Anti-CCP2 Status [Number; unit: participants] — Anti-citrullinated protein/peptide antibodies (ACPA) are among the most disease-specific autoantibodies for rheumatoid arthritis (RA). These antibodies occur specifically in RA and can be measured most conveniently via the anti-CCP (anti-cyclic citrullinated peptide) antibody test. The anti-CCP2 test enables clinicians to distinguish RA patients from other arthritic diseases, especially in cases where the RF test is not discriminative.
  participants
    Negative | 14 | 6 | 20
    Positive | 13 | 17 | 30
Duration of Rheumatoid Arthritis [Mean (Standard Deviation); unit: months] | 25.7 (18.0) | 28.2 (17.0) | 26.8 (17.4)
Disease Activity Score (DAS) 28 (C-Reactive Protein [CRP]) [Mean (Standard Deviation); unit: units on a scale] — The DAS28 is a continuous disease measure which is a composite of 4 variables: the 28 tender joint count, the 28 swollen joint count, CRP, and participant assessment of disease activity measure on a visual analogue scale. The DAS28 has numeric thresholds that define high disease activity (> 5.1), low disease activity (< 3.2) and remission (< 2.6). A clinically significant response= decrease in DAS28 score of >1.2 from baseline. DAS28 area under the curve (DAS28AUC) can be calculated from the DAS28 score versus time curve, which provides an assessment of changes in disease activity over time.
  units on a scale | 5.3 (1.1) | 5.3 (0.9) | 5.3 (1.0)
Number of Tender Joints [Mean (Standard Deviation); unit: joints] | 12.9 (7.1) | 13.3 (7.2) | 13.1 (7.2)
Number of Swollen Joints [Mean (Standard Deviation); unit: joints] | 11.3 (6.6) | 8.5 (4.1) | 10.0 (5.7)
Cross Classification of RF Status and CCP2 Status at Baseline [Number; unit: participants] — Venous blood was collected and tested for rheumatoid factor and anti-CCP antibodies. RF was measured by an immunoturbidimetric assay (Roche Tina-Quant). Anti-CCP was measured by an anti-CCP2 immunoassay.
  participants
    RF negative, anti-CCP2 negative | 12 | 3 | 15
    RF negative, anti-CCP2 positive | 0 | 1 | 1
    RF positive, anti-CCP2 negative | 2 | 3 | 5
    RF positive, anti-CCP2 positive | 13 | 16 | 29

OUTCOME MEASURES:

1. Primary Outcome: Double-blind Period: Mean Synovitis Scores at Baseline As Measured by the Rheumatoid Arthritis Clinical Trials 6 (OMERACT 6) Rheumatoid Arthritis Magnetic Resonance Imaging Score (RAMRIS)
Description: Wrist synovitis was assessed by postgadolinium MRI enhancement according to OMERACT 6 RAMRIS in 3 wrist regions: distal radioulnar, radiocarpal, and intercarpal and carpometacarpal joints. For each wrist region, possible score ranges from 0-3, with 0=normal, 1=mild, 2=moderate, and 3=severe damage. The total synovitis score per wrist=the sum of the individual scores for the 3 wrist regions. Minimum score per wrist ranges from 0, indicating no damage, to 9 (score of 3*3 wrist regions), indicating most severe damage. Change in synovitis = Follow-up synovitis score - baseline score.
Time Frame: At baseline
Population: All randomized participants who received at least 1 dose of study medication and had synovitis assessments available at baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Abatacept + Methotrexate: Abatacept was administered intravenously on Days 1, 15, and 29 and every 28 days up to and including Day 113. Abatacept dose was based on body weight: 500 mg for participants weighing <60 kg, 750 mg for participants weighing 60 to 100 kg, and 1 gram for participants weighing >100 kg.
- Placebo + Methotrexate: Placebo was administered IV on Days 1, 15, and 29 and every 28 days up to and including Day 113. In addition, participants received a weekly dose of at least 15 mg (or a maximum tolerated dose, such as 10 mg weekly) of methotrexate).
Arm/Group | Abatacept + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 25 | 23
units on a scale | 4.48 (2.10) | 3.52 (2.43)

2. Secondary Outcome: Double-blind Period: Baseline Mean Erosion OMERACT 6 Scores
Description: Bone erosion assessed at a total of 23 anatomic locations: 15 in 1 wrist and 8 in the hand of the same side. Each site is scored in 1.0 increments from 0 (no damage) to 10 (severe damage) according to erosion of the original articular bone (each unit=10% loss of articular bone). The total erosion score for the hands/wrists is the sum of the individual scores for each location. Thus the maximum score achievable per hand/wrist is 230. Increasing score=greater severity.
Time Frame: At baseline
Population: All randomized participants who received at least 1 dose of study medication and had erosion OMERACT 6 assessments available at baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo + Methotrexate: Placebo was administered IV on Days 1, 15, and 29 and every 28 days up to and including Day 113. In addition, participants received a weekly dose of at least 15 mg (or a maximum tolerated dose, such as 10 mg weekly) of methotrexate.
Arm/Group | Abatacept + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 25 | 23
units on a scale | 12.60 (9.41) | 9.65 (10.11)

3. Secondary Outcome: Double-blind Period: Adjusted Mean Change From Baseline in Erosion OMERACT 6 Scores
Description: Bone erosion assessed at 23 anatomic locations: 15 in 1 wrist and 8 in attached hand. Each site is scored in 1.0 increments from 0 (no damage) to 10 (severe damage), indicating erosion (each unit=10% bone loss) of original articular bone. Total erosion score for hands/wrists is sum of the individual scores for each location. Thus the maximum score per hand/wrist is 230. Increasing score=greater severity. Adjusted change from baseline in erosion score=mean score at Day 113-mean erosion score at baseline. Adjustment based on ANCOVA model with treatment=factor and baseline value=covariate.
Time Frame: Baseline to Day 113
Population: All randomized participants who received at least 1 dose of study medication and had erosion OMERACT 6 assessments available at baseline and Day 113.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Abatacept + Methotrexate: Abatacept was administered IV and including Day 113. Abatacept dose was based on body weight: 500 mg for participants weighing <60 kg, 750 mg for participants weighing 60 to 100 kg, and 1 gram for participants weighing >100 kg.
Arm/Group | Abatacept + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 25 | 23
units on a scale | 0.45 (0.43) | 0.95 (0.45)
Statistical Analysis 1: Comparison: Abatacept + Methotrexate vs Placebo + Methotrexate; Comparison in the change from baseline of erosion score using the OMERACT 6 RA MRI score method between Abatacept and Placebo at Day 113 was based on a non-parametric analysis of covariance model (ANCOVA). Change from BL = Post-BL measurement-BL value. Adjustment was based on ANCOVA model with treatment as a factor and BL value a covariate; Test type: Superiority or Other; ANCOVA; Adjusted Mean Difference from Placebo = -0.50, 95% CI 2-sided [-1.77 to 0.76]

4. Primary Outcome: Double-blind Period: Mean Change From Baseline in OMERACT 6 Wrist Synovitis Score: Planned Analysis Using Non-Parametric ANCOVA
Description: Wrist synovitis was assessed by postgadolinium MRI enhancement according to OMERACT 6 RAMRIS in 3 wrist regions: distal radioulnar, radiocarpal, and intercarpal and carpometacarpal joints. For each wrist region, possible score ranges from 0-3, with 0=normal, 1=mild, 2=moderate, and 3=severe damage. The total synovitis score per wrist=the sum of the individual scores for the 3 wrist regions. Minimum score per wrist ranges from 0, indicating no damage, to 9 (score of 3*3 wrist regions), indicating most severe damage. Change in synovitis=Follow-up synovitis score-baseline score.
Time Frame: Baseline to Day 113
Population: All randomized participants who received at least 1 dose of study medication and had wrist synovitis assessments available at baseline and Day 113.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Abatacept + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 25 | 23
units on a scale | -0.44 (1.47) | 0.52 (1.38)
Statistical Analysis 1: Comparison: Abatacept + Methotrexate vs Placebo + Methotrexate; Comparison in change from baseline of wrist synovitis using OMERACT 6 rheumatoid arthritis magnetic resonance imaging score method between abatacept and placebo at Day 113 based on a nonparametric analysis of covariance model. Baseline and changes from baseline of the total wrist synovitis scores were ranked, and the model included the rank score for change from baseline as the dependent variable with treatment group as a main effect and the rank score for baseline as an additional covariate; Test type: Superiority or Other; p = 0.103, ANCOVA; Mean Difference (Final Values) = 0.96

5. Secondary Outcome: Double-blind Period: Baseline Mean Osteitis OMERACT 6 Scores
Description: Osteitis assessed at a total of 23 anatomic locations: 15 in 1 wrist and 8 in the hand of the same side. Each site is scored in 1.0 increments from 0 to 3, indicating involvement of original articular bone. The total score for the hands/wrists is the sum of the individual scores for each location. Thus the maximum score achievable per hand/wrist is 23 (total number of anatomic locations) * 3 (maximum per joint)=69. Minimum score=0, indicating normal. Increasing score=greater severity.
Time Frame: At baseline
Population: All randomized participants who received at least 1 dose of study medication and had osteitis OMERACT 6 assessments available at baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Abatacept + Methotrexate: Abatacept was administered IV on Days 1, 15, and 29 and every 28 days up to and including Day 113. Abatacept dose was based on body weight: 500 mg for participants weighing <60 kg, 750 mg for participants weighing 60 to 100 kg, and 1 gram for participants weighing >100 kg.
Arm/Group | Abatacept + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 25 | 23
units on a scale | 7.72 (7.04) | 8.00 (9.72)

6. Secondary Outcome: Double-blind Period: Adjusted Mean Change From Baseline in Osteitis OMERACT 6 Scores
Description: Osteitis assessed at 23 anatomic locations: 15 in 1 wrist and 8 in attached. Each site scored in 1.0 increments, indicating involvement of original articular bone (0=none to 3=severe). Total score for hands/wrists is sum of scores for each location. Maximum score per hand/wrist is 23 (total anatomic locations)*3 (maximum score per joint)=69. Minimum score=0(normal). Increasing score=greater severity. Adjusted mean change from baseline in osteitis score=mean score at Day 113-mean score at baseline. Adjustment based on ANCOVA model with treatment=factor and baseline value=covariate.
Time Frame: Baseline to Day 113
Population: All randomized participants who received at least 1 dose of study medication and had osteitis OMERACT 6 assessments available at baseline and Day 113.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Abatacept + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 25 | 23
units on a scale | -1.94 (0.86) | 1.54 (0.90)
Statistical Analysis 1: Comparison: Abatacept + Methotrexate vs Placebo + Methotrexate; Comparison in the change from baseline of Edema/Osteitis score using the OMERACT 6 RA MRI score method between Abatacept and Placebo at Day 113 was based on a non-parametric analysis of covariance model (ANCOVA). Change from BL = Post-BL measurement-BL value. Adjustment was based on ANCOVA model with treatment as a factor and BL value a covariate; Test type: Superiority or Other; ANCOVA; Adjusted Mean Difference from Placebo = -3.48, 95% CI 2-sided [-6.00 to -0.96]

7. Secondary Outcome: Double-blind Period: Number of Participants With Newly Involved Joints in Bone Erosion, Edema/Osteitis, and Synovitis
Description: Bone erosion and osteitis were assessed at a total of 23 anatomic locations according to erosion (for bone erosion) or involvement (for osteitis) of the original articular bone. Synovitis assessed as above-normal post-gadolinium enhancement in 3 wrist regions: distal radioulnar joint, radiocarpal joint, and intercarpal and carpometacarpal joints.
Time Frame: Baseline to Day 113
Population: All randomized participants who received at least 1 dose of study medication and had erosion, edema, and synovitis assessments available at baseline and Day 113.
Measure: Number; unit: participants
Arm/Group | Abatacept + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 25 | 23
participants
  0 newly involved joints (Bone Erosion) | 20 | 16
  ≥1 newly involved joints (Bone Erosion) | 5 | 7
  0 newly involved joints (Edema/Osteitis) | 18 | 16
  ≥1 newly involved joints (Edema/Osteitis) | 7 | 7
  0 newly involved joints (Synovitis) | 23 | 20
  ≥1 newly involved joints (Synovitis) | 2 | 3

8. Secondary Outcome: Double-blind Period: Baseline Mean RAMRIS Scores
Description: RAMRIS score is the sum of its core components: Synovitis Score, Osteitis Score, and Erosion Score. Synovitis scored from 0 (normal) to 9 (maximum distension of synovial cavity). Osteitis scored 0 (normal) to 69 (maximum articular bone involvement). Erosion scored from 0 (normal) to 230 (maximum erosion of articular bone). RAMRIS=Synovial Score + Osteitis Score + Erosion Score. Minimum RAMRIS score=0 (normal), maximum RAMRIS score=308 (severe structural damage). For Synovial Score, Osteitis Score, Erosion Score, and RAMRIS score, increasing number=increasing severity.
Time Frame: Baseline
Population: All randomized participants who received at least 1 dose of study medication and had RAMRIS assessments available at baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Abatacept + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 25 | 23
units on a scale | 24.80 (16.36) | 21.17 (20.45)

9. Secondary Outcome: Double-blind Period: Adjusted Mean Change From Baseline in RAMRIS Scores
Description: RAMRIS Score=sum of core components: Synovitis (S), Osteitis (O), and Erosion (E) Scores. S scored 0 (none) to 9 (maximum distension of synovial cavity); O scored 0 (none) to 69 (maximum articular bone involvement); E scored 0 (none) to 230 (maximum erosion of articular bone). RAMRIS=S+O+E Scores. RAMRIS minimum score=0 (normal), maximum=308 (severe structural damage). Adjusted change from baseline in RAMRIS=mean RAMRIS at Day 113-mean RAMRIS at baseline. Adjustment based on ANCOVA model: treatment=factor, baseline value=covariate.
Time Frame: Baseline to Day 113
Population: All randomized participants who received at least 1 dose of study medication and had RAMRIS assessments available at baseline and Day 113.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Abatacept + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 25 | 23
units on a scale | -1.82 (1.13) | 2.89 (1.18)
Statistical Analysis 1: Comparison: Abatacept + Methotrexate vs Placebo + Methotrexate; Comparison in the change from baseline of RAMRIS score using the OMERACT 6 RA MRI score method between Abatacept and Placebo at Day 113 was based on a non-parametric analysis of covariance model (ANCOVA). Change from BL = Post-BL measurement-BL value. Adjustment was based on ANCOVA model with treatment as a factor and BL value a covariate; Test type: Superiority or Other; ANCOVA; Adjusted Mean Difference from Placebo = -4.71, 95% CI 2-sided [-8.00 to -1.42]

10. Secondary Outcome: Double-blind Period: Median Percent Change From Baseline in Systemic Markers of Bone Formation: Osteocalcin and Serum Intact N-terminal Propeptide of Type I Procollagen (PINP)
Description: PINP and osteocalcin are markers of bone formation. Osteocalcin is synthesized by osteoblasts and is associated with osteoblast synthetic activity. Osteoblasts secrete type 1 procollagen, and cleavage of large fragments from the carboxy and amino terminal ends result in formation of mature type 1 collagen and production of PINP fragments.
Time Frame: Baseline to Days 15, 29, 57, 85, and 113
Population: All randomized participants who received at least 1 dose of study medication.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Abatacept + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 27 | 23
percent change
  Day 15 osteocalcin (n=25, n=21) | 1.82 [-10.2 to 12.1] | 4.41 [-12.7 to 15.6]
  Day 15 serum intact PINP (n=25, n=21) | 6.83 [-3.9 to 15.7] | 3.94 [-8.4 to 13.9]
  Day 29 osteocalcin (n=26, n=21) | 2.43 [-8.8 to 18.2] | 12.14 [-10.1 to 19.2]
  Day 29 serum intact PINP (n=26, n=21) | 11.62 [1.1 to 30.8] | -0.18 [-9.3 to 23.5]
  Day 57 osteocalcin (n=25, n=21) | 4.02 [-7.7 to 25.4] | 10.53 [-3.7 to 22.8]
  Day 57 serum intact PINP (n=25, n=21) | 3.68 [-8.1 to 43.1] | 12.18 [-6.7 to 20.2]
  Day 85 osteocalcin (n=24, n=21) | 4.76 [-11.5 to 34.1] | 10.62 [-14.8 to 25.8]
  Day 85 serum intact PINP (n=24, n=21) | 5.97 [-10.6 to 36.3] | -7.23 [-18.1 to 14.8]
  Day 113 osteocalcin (n=24, n=21) | 3.18 [-8.2 to 11.8] | 7.87 [-8.3 to 19.0]
  Day 113 serum intact PINP (n=24, n=21) | 2.98 [-19.8 to 28.8] | 4.75 [-16.1 to 24.7]

11. Secondary Outcome: Double-blind Period: Median Percent Change From Baseline in Systemic Markers of Bone Destruction (Serum Carboxy-terminal Cross-linking Telopeptide of Type I Collagen [CTX-I] and Serum Pyridinoline Cross-linked Telopeptide Domain of Type I Collagen [ICTP])
Description: CTX-I and ICTP are biochemical markers of bone resorption or bone degradation
Time Frame: Baseline to Days 15, 29, 57, 85, and 113
Population: All randomized participants who received at least 1 dose of study medication.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Abatacept + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 27 | 23
percent change
  Day 15 CTX-1 (n=25, n=21) | 1.65 [-23.0 to 13.0] | -6.37 [-24.6 to 23.2]
  Day 15 ICTP (n=25, n=21) | -5.56 [-17.1 to 10.9] | 6.25 [-6.2 to 18.6]
  Day 29 CTX-1 (n=26, n=21) | 0.48 [-28.2 to 32.2] | -0.72 [-21.2 to 18.6]
  Day 29 ICTP (n=26, n=21) | -3.47 [-10.1 to 10.0] | 4.34 [-3.7 to 20.4]
  Day 57 CTX-1 (n=25, n=21) | 15.13 [-17.9 to 26.5] | 7.02 [-11.4 to 16.7]
  Day 57 ICTP (n=25, n=21) | -5.08 [-15.9 to 14.5] | 8.73 [-3.7 to 21.6]
  Day 85 CTX-1 (n=24, n=21) | -6.94 [-35.9 to 21.5] | 15.65 [-18.9 to 40.8]
  Day 85 ICTP (n=24, n=21) | -6.36 [-24.7 to 4.7] | 2.25 [-7.1 to 9.7]
  Day 113 CTX-1 (n=24, n=21) | -7.23 [-36.4 to 21.3] | 0.00 [-27.5 to 35.3]
  Day 113 ICTP (n=24, n=21) | -11.29 [-27.7 to 1.5] | 11.64 [-2.2 to 29.9]

12. Secondary Outcome: Double-blind Period: Median Percent Change From Baseline in a Systemic Marker of Cartilage Degradation (Creatinine-corrected Urinary Carboxyterminal Crosslinking Telopeptide of Type II Collagen [UCTX2C])
Description: Urinary CTX-II is a biochemical marker of type II collagen breakdown. In participants with early rheumatoid arthritis, increased levels of CTX-II can be predictive of rapid radiographic progression over periods of 1 to 5 years. These markers of cartilage destruction can predict progression of joint damage, independent of clinical and biologic indices of disease activity and baseline joint damage.
Time Frame: Baseline to Days 15, 29, 57, 85, and 113
Population: All randomized participants who received at least 1 dose of study medication.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Abatacept + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 27 | 23
percent change
  Day 15 UCTX2C (n=24, n=21) | -8.51 [-35.9 to 13.7] | 5.14 [-11.7 to 8.4]
  Day 29 UCTX2C (n=21, n=19) | -3.40 [-16.5 to 5.8] | 6.81 [-25.1 to 13.5]
  Day 57 UCTX2C (n=23, n=19) | 0.24 [-50.0 to 25.0] | 5.43 [-12.3 to 24.8]
  Day 85 UCTX2C (n=22, n=20) | -10.83 [-38.4 to 14.7] | 9.67 [-13.8 to 29.2]
  Day 113 UCTX2C (n=22, n=20) | -18.49 [-46.9 to 54.2] | 9.86 [-22.4 to 46.3]

13. Secondary Outcome: Double-blind Period: Median Percent Change From Baseline in Systemic Marker of Synovial Tissue Metabolism (Creatinine-corrected Urinary Glucosyl-Galactosyl-Pyridinoline [UGGPC])
Description: Glucosyl-galactosyl-pyridinoline (Glc-Gal-PYD) is a specific biochemical marker reflecting the degradation of the synovial tissue membrane. It is a glycosylated derivative of the collagen crosslink pyridinoline, and it is present in significant amounts only in the synovial membrane; it is absent from bone and present in minutes amounts in cartilage and other soft tissues. Increased urinary levels of Glc-Gal-PYD have been found in early and long-standing rheumatoid arthritis, high levels being associated with rapid destruction.
Time Frame: Baseline to Days 15, 29, 57, 85, and 113
Population: All randomized participants who received at least 1 dose of study medication.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Abatacept + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 27 | 23
percent change
  Day 15 UGGPC (n=24, n=20) | 4.44 [-20.5 to 65.0] | -3.84 [-13.7 to 12.4]
  Day 29 UGGPC (n=22, n=18) | -1.83 [-19.3 to 76.9] | -3.19 [-25.6 to 26.8]
  Day 57 UGGPC (n=23, n=16) | 1.58 [-24.8 to 23.4] | 5.73 [-12.6 to 28.2]
  Day 85 UGGPC (n=22, n=18) | 0.32 [-31.0 to 54.5] | 16.29 [-14.4 to 39.7]
  Day 113 UGGPC (n=22, n=18) | -12.16 [-27.9 to 53.3] | -3.10 [-31.5 to 32.3]

14. Secondary Outcome: Double-blind Period: Number of Participants With Death, Serious Adverse Events (SAEs), Treatment-related SAEs, SAEs Leading to Discontinuation, Adverse Events (AEs), Treatment-related AEs, and AEs Leading to Discontinuation
Description: An AE is any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that does not necessarily have a causal relationship with treatment. An SAE is any unfavorable medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency or abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Treatment-related=possibly, probably, or certainly related to and of unknown relationship to study treatment.
Time Frame: From Day 1 to Day 113, and up to 56 days post last dose of double-blind period, or start of first dose of open-label period
Population: All randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Abatacept + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 27 | 23
participants
  Deaths | 0 | 0
  SAEs | 0 | 2
  Treatment-related SAEs | 0 | 0
  SAEs Leading to Discontinuation | 0 | 0
  AEs | 20 | 14
  Treatment-related AEs | 8 | 6
  AEs Leading to Discontinuation | 0 | 0

15. Secondary Outcome: Double-blind Period: Number of Participants With AEs of Special Interest
Description: An AE is any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that does not necessarily have a causal relationship with treatment. AEs of special interest are those AEs that may be associated with the use of immunomodulatory drugs, including serious, opportunistic, and all other infections; autoimmune disorders; neoplasms; acute infusional AEs (prespecified AEs occurring within 1 hour of start of infusion) and peri-infusional AEs (prespecified AEs occurring within 24 hours of start of infusion).
Time Frame: as for outcome 14
Population: All randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Abatacept + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 27 | 23
participants
  Infections | 1 | 0
  Malignancies | 0 | 0
  Autoimmune disorders | 0 | 0
  Acute infusional AEs | 0 | 4
  Peri-infusional AEs | 4 | 5

16. Secondary Outcome: Double-blind Period: Number of Participants With Infections/Infestations of Special Interest
Description: Infections/Infestations of Special Interest are AEs and SAEs considered possibly, probably, or certainly related to study treatment, graded according to Common Terminology Criteria for Adverse Events Version 3.0 (Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe, Grade 4=Life-threatening or disabling, Grade 5=Death). AE=any new untoward medical occurrence or worsening of a preexisting medical condition which does not necessarily have a causal relationship with this treatment.
Time Frame: as for outcome 14
Population: All randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Abatacept + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 27 | 23
participants | 1 | 0

17. Secondary Outcome: Double-blind Period: Number of Participants With Acute Infusional AEs of Special Interest
Description: Acute infusional AEs are AEs with onset during the first hour after the start of study drug infusion. An AE is any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that does not necessarily have a causal relationship with treatment. AEs considered possibly, probably, or certainly related to study treatment were graded according to Common Terminology Criteria for Adverse Events ,Version 3.0 (Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe, Grade 4=Life-threatening or disabling, Grade 5=Death).
Time Frame: as for outcome 14
Population: All randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Groups:
- Placebo (PLA) + MTX: Placebo was administered IV on Days 1, 15, and 29 and every 28 days up to and including Day 113. In addition, participants received a weekly dose of at least 15 mg (or a maximum tolerated dose, such as 10 mg weekly) of methotrexate.
Arm/Group | Abatacept + Methotrexate | Placebo (PLA) + MTX
Number analyzed (Participants) | 27 | 23
participants
  Grade 1 diarrhea | 0 | 1
  Grade 1 overdose | 0 | 1
  Grade 1 headache | 0 | 1
  Grade 1 flushing | 0 | 1

18. Secondary Outcome: Double-blind Period: Number of Participants With Peri-infusional AEs of Special Interest
Description: Peri-infusional AEs are AEs occurring during the first 24 hours after the start of study drug infusion. An AE is any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that does not necessarily have a causal relationship with treatment. AEs considered possibly, probably, or certainly related to study treatment were graded according to Common Terminology Criteria for Adverse Events, Version 3.0 (Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe, Grade 4=Life-threatening or disabling, Grade 5=Death).
Time Frame: as for outcome 14
Population: All randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Abatacept + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 27 | 23
participants
  Grade 1 nausea | 3 | 0
  Grade 1 headache | 0 | 1
  Grade 2 headache | 1 | 1
  Grade 1 flushing | 0 | 2
  Grade 2 arthralgia | 0 | 1
  Grade 1 cough | 0 | 1

19. Secondary Outcome: Double-blind Period: Number of Participants With Laboratory Test Results in Hematology Meeting the Criteria for Marked Abnormality
Description: BL=baseline; LLN=lower limit of normal; ULN=upper limit of normal. Marked abnormality criteria: Hemoglobin: >3 g/dL decrease from BL. Hematocrit: <0.75*BL. Erythrocytes: <0.75*BL. Platelets: <0.67*LLN/>1.5*ULN, or if BL <LLN, use 0.5*BL/<100,000 mm^3. Leukocytes: <0.75*LLN/>1.25*ULN, or if BL<LLN, use <0.8*BL/>ULN, or if BL>ULN, use >1.2*BL/<LLN. Neutrophils+bands: <1.0*10^3 c/uL. Eosinophils: >0.750*10^3 c/uL. Basophils: > 400 mm^3. Monocytes: >2000 mm^3. Lymphocytes: <0.750*10^3 c/uL/>7.50*10^3 c/uL.
Time Frame: as for outcome 14
Population: All randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Abatacept + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 27 | 23
participants
  Low hemoglobin | 0 | 1
  Low hematocrit | 0 | 1
  Low erythrocytes | 0 | 0
  Low platelets | 0 | 0
  High platelets | 0 | 1
  Low leukocytes | 0 | 0
  High leukocytes | 1 | 0
  Low neutrophils+bands | 0 | 1
  Low lymphocytes | 2 | 2
  High lymphocytes | 0 | 0
  High monocytes | 0 | 0
  High basophils | 0 | 0
  High eosinophils | 0 | 0

20. Secondary Outcome: Double-blind Period: Number of Participants With Laboratory Test Results for Liver and Kidney Function Meeting Criteria for Marked Abnormality
Description: ULN=upper limit of normal; BL=baseline. Marked abnormality criteria: Alkaline phosphatase: >2*ULN, or if BL>ULN, use >3*BL; aspartate aminotransferase: >3*ULN, or if BL>ULN,use >4*BL; alanine aminotransferase: >3*ULN, or if BL>ULN, use >4*BL; G-Glutamyl transferase: >2*ULN, or if BL>ULN, use >3*BL; Bilirubin: >2*ULN, or if BL>ULN, use >4*BL; blood urea nitrogen: >2*BL; creatinine: >1.5*BL.
Time Frame: From Day 1 to Day 113, and including up to 56 days post last dose of double-blind period, or start of first dose of open-label period
Population: All randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Abatacept + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 27 | 23
participants
  High alkaline phosphatase | 0 | 0
  High aspartate aminotransferase | 0 | 0
  High alanine aminotransferase | 0 | 0
  High G-Glutamyl transferase | 0 | 0
  High bilirubin | 0 | 0
  High blood urea nitrogen | 0 | 0
  High creatinine | 1 | 0

21. Secondary Outcome: Double-blind Period: Number of Participants With Laboratory Test Results for Electrolytes Meeting the Criteria for Marked Abnormality
Description: LLN=lower limit of normal; ULN=upper limit of normal; BL=baseline. Marked abnormality: Sodium: <0.95*LLN/>1.05*ULN,or if BL<LLN, use 0.95*BL or >ULN,or if BL>ULN, use>1.05*BL or <LLN. Potassium: <0.9*LLN/>1.1* ULN,or if BL<LLN, use 0.9*BL or >ULN, or if BL>ULN, use>1.1*BL or <LLN. Chloride: <0.9*LLN/>1.1*ULN, or if BL<LLN, use 0.9*BL or >ULN, or if BL>ULN, use>1.1*BL or <LLN. Calcium: <0.8*LLN/>1.2*ULN, or if BL<LLN, use 0.75*BL or >ULN, or if BL>ULN, use>1.25*BL or <LLN. Phosphorous: <0.75*LLN/>1.25*ULN, or if BL<LLN, use 0.67*BL or >ULN, or if BL>ULN, use>1.33*BL or <LLN.
Time Frame: as for outcome 14
Population: All randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Abatacept + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 27 | 23
participants
  Low sodium | 0 | 0
  High sodium | 0 | 0
  Low potassium | 0 | 0
  High potassium | 1 | 0
  Low chloride | 0 | 0
  High chloride | 0 | 0
  Low calcium | 0 | 0
  High calcium | 0 | 0
  Low phosphorous | 0 | 0
  High phosphorous | 0 | 0

22. Secondary Outcome: Double-blind Period: Number of Participants With Laboratory Test Results in Other Chemistries and Urinalysis Meeting the Criteria for Marked Abnormality
Description: LLN=lower limit of normal; ULN=upper limit of normal; BL-baseline. Marked abnormality c: serum glucose:<65 mg/dL/>220 mg/dL; fasting serum glucose: <0.8* LLN/>1.5* ULN, or if BL<LLN, use 0.8*BL or >ULN, or if BL>ULN, use >2.0*BL or <LLN; total protein: <0.9*LLN/>1.1* ULN; albumin: <0.9*LLN,or if BL<LLN, use <0.75 BL; uric acid: >1.5* ULN, or if BL>ULN, use >2*BL. Urinalysis (Urine protein, urine Glu, urine blood, leukocyte esterase, red blood cells, white blood cells):Use ≥2 when BL value missing or value ≥4,or when predose=0 or 0.5. Use ≥3 when predose=1. Use ≥4 when predose=2 or 3
Time Frame: as for outcome 14
Population: All randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Abatacept + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 27 | 23
participants
  Low serum glucose (n=27, n=23) | 1 | 0
  High serum glucose (n=27, n=23) | 1 | 1
  Low fasting glucose (n=20, n=17) | 0 | 0
  High fasting glucose (n=20, n=17) | 1 | 0
  Low total protein (n=27, n=23) | 0 | 0
  High total protein (n=27, n=23) | 0 | 0
  Low albumin (n=27, n=23) | 0 | 0
  High uric acid (n=27, n=23) | 0 | 0
  High urine protein (n=27, n=23) | 1 | 1
  High urine glucose (n=27, n=23) | 0 | 0
  High urine blood (n=27, n=23) | 2 | 1
  High leukocyte esterase (n=27, n=23) | 4 | 4
  High urine white blood cells (n=10, n=9) | 2 | 3
  High urine red blood cells (n=10, n=8) | 3 | 3

23. Primary Outcome: Double-blind Period: Mean Change From Baseline in OMERACT 6 Wrist Synovitis Score: Post Hoc Sensitivity Analysis Using Parametric ANCOVA Analysis
Description: Wrist synovitis was assessed by postgadolinium MRI enhancement according to OMERACT 6 RAMRIS in 3 wrist regions: distal radioulnar, radiocarpal, and intercarpal and carpometacarpal joints. For each wrist region, possible score ranges from 0-3, with 0=normal, 1=mild, 2=moderate, and 3=severe damage. The total synovitis score per wrist=the sum of the individual scores for the 3 wrist regions. Minimum score per wrist ranges from 0, indicating no damage, to 9 (score of 3*3 wrist regions), indicating most severe damage. Change in synovitis score=Follow-up synovitis score-baseline synovitis score.
Time Frame: Baseline to Day 113
Population: All randomized participants who received at least 1 dose of study medication and who had wrist synovitis assessments available at baseline and Day 113.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo (PLA) + MTX: Placebo was administered IV on Days 1, 15, and 29 and every 28 days up to and including Day 113. In addition, participants received a weekly dose of at least 15 mg (or a maximum tolerated dose, such as 10 mg weekly) of methotrexate).
Arm/Group | Abatacept + Methotrexate | Placebo (PLA) + MTX
Number analyzed (Participants) | 25 | 23
units on a scale | -0.31 (0.26) | 0.38 (0.27)
Statistical Analysis 1: Comparison: Abatacept + Methotrexate vs Placebo (PLA) + MTX; Comparison in change from baseline of wrist synovitis using OMERACT 6 rheumatoid arthritis magnetic resonance imaging (MRI) score method between ABA and PLA at Day 113 based on a parametric analysis of covariance model (ANCOVA). The model included the score change from baseline as the dependent variable, treatment group as a main effect and baseline score as an additional covariate; Test type: Superiority or Other; p = 0.078, ANCOVA; Mean Difference (Net) = 0.69

24. Secondary Outcome: Double-blind Period:Number of Participants With Significantly Abnormal Changes in Vital Signs
Description: Vital signs, which included blood pressure, heart rate, respiration, and temperature, were monitored predose and 1 hour after start of infusion. Changes in vital signs were determined to be significantly abnormal at the discretion of the investigator but were generally those that either exceeded, or failed to reach, normal parameters. Normal vital sign parameter ranges varied by site.
Time Frame: Days 1, 15, 29, 57, 85, and 113
Population: All randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Abatacept + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 27 | 23
participants | 0 | 0

25. Secondary Outcome: Double-blind Period: Number of Participants With Positive Antibodies to Abatacept by Electrochemiluminescence (ECL) Assay
Description: On-Rx=on treatment; post-Rx=post treatment. ECL screened sera for drug-specific antibodies; immunocompetition was used to identify specific anti-Abatacept reactivity. Cytotoxic leukocyte antigen 4 (CTLA4) and Possibly Immunoglobulin (Ig) Category=reactivity against extracellular domain of human CTLA4, constant regions of human IgG1, or both (CTLA4Ig; Abatacept molecule). Ig and/or Junction Category=reactivity against constant regions and/or hinge region of human IgG1.
Time Frame: Day 1 to Day 113
Population: All randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Abatacept + Methotrexate
Number analyzed (Participants) | 27
participants
  Overall on-Rx visits, CTLA4 + possibly Ig (n=27) | 0
  Overall on-Rx visits, Ig and/or junction (n=27) | 0
  Overall post-Rx visits, CTLA4 + possibly Ig (n=1) | 0
  Overall post-Rx visits, Ig and/or junction (n=1) | 0
  Overall visits, CTLA4 + possibly Ig (n=27) | 0
  Overall visits, Ig and/or junction (n=27) | 0

ADVERSE EVENTS:
Groups:
- ABA + MTX: Abatacept was administered IV on Day 1, 15, 29 and every 28 days up to and including Day 113.Abatacept was given as a dose based on body weight: 500 mg for participants weighing < 60 kg, 750 mg for participants weighing 60 to 100 kg and 1 gram for participants weighing > 100 kg. In addition, participants received a weekly dose of MTX of at least 15 mg or a maximum tolerated dose (ie, 10 mg weekly)
- PLA + MTX: PLA was administered IV on Day 1, 15, 29 and every 28 days up to and including Day 113. In addition, participants received a weekly dose of MTX of at least 15 mg or a maximum tolerated dose (ie, 10 mg weekly)
Arm/Group | ABA + MTX | PLA + MTX
Serious Adverse Events (participants affected / at risk) | 0/27 | 2/23
Other Adverse Events (participants affected / at risk) | 12/27 | 8/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABA + MTX (N=27) | PLA + MTX (N=23)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 1
OVERDOSE (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ABA + MTX (N=27) | PLA + MTX (N=23)
FLUSHING (Vascular disorders) | 0 | 2
HEADACHE (Nervous system disorders) | 1 | 2
DIZZINESS (Nervous system disorders) | 2 | 0
NAUSEA (Gastrointestinal disorders) | 4 | 0
DIARRHOEA (Gastrointestinal disorders) | 2 | 1
SINUSITIS (Infections and infestations) | 2 | 0
NASOPHARYNGITIS (Infections and infestations) | 1 | 2
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 2
FATIGUE (General disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.